CLINICAL TRIAL: NCT06623760
Title: Intervention Study：Study on the Impact of Desk and Chair Adaptation Intervention on the Occurrence and Development of Myopia in Primary School Students
Brief Title: Study on the Impact of Desk and Chair Adaptation Intervention on the Occurrence and Development of Myopia in Primary School Students
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fangbiao Tao (Other)
Responsible Party: Sponsor-Investigator, Fangbiao Tao, Professor, Anhui Medical University
Organization: Anhui Medical University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 20240901
Record Dates: First submitted 2024-09-30; First posted 2024-10-02 (Actual); Last update posted 2024-10-02 (Actual); Status verified 2024-08

CONDITIONS: Axial Length, Eye; Myopia; Myopia Progression
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Desk and chair adaptation interventions (Experimental): Adjustment of the height of desks and chairs according to the height of each student, intervention lasting one year
  Interventions: Device: Desk and chair adaptation interventions
- Continued use of original desks and chairs (No Intervention): No change in height of desks and chairs, use as usual

INTERVENTIONS:
Device: Desk and chair adaptation interventions — Adjustment of the height of tables and chairs to the height of each pupil in accordance with Functional sizes and technical requirements of chairs and tables for educational institutions (GB/T 3976--2014）, with a duration of intervention of one year。
  Arms: Desk and chair adaptation interventions

SUMMARY:
This study is a randomized controlled trial of a desk and chair adaptation intervention involving primary school students and their parents or primary caregivers. We compared the myopia status of students in the intervention and control groups before and after the intervention to confirm the effect of the desk and chair adaptation intervention on the development of myopia in students.

DETAILED DESCRIPTION:
In this study, two pilot schools in Anhui Province were selected , and all students were examined by ophthalmologists, and their heights and the heights of their desks and chairs were measured in order to investigate the association between desk and chair adaptations and myopia. One of the elementary school was randomly selected for a one-year desk and chair adaptation intervention to compare the occurrence of myopia and axial growth of the students before and after the intervention in the two schools.

Translated with DeepL.com (free version)

ELIGIBILITY:
Inclusion Criteria:

* Students and their families were informed and voluntarily participated in the study, with parents signing the informed consent form.
* Able to cooperate with eye examinations and questionnaires.

Exclusion Criteria:

* Communication barriers, unable to cooperate.
* Strabismus, amblyopia, or any other ocular or systemic diseases that may affect refractive development.
* Children currently using orthokeratology lenses or rigid contact lenses.
* Using other interventions (such as acupuncture, massage, medication, ear acupuncture, etc.) to control myopia, apart from school eye exercises.

Ages: 6 Years to 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 2100 (Estimated)
Dates: Start 2024-10-01 (Estimated); Primary Completion 2025-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
The changes in axial length (AL) and spherical equivalent (SE) compared to baseline after one year of intervention | at baseline, , and at the 12th month of the intervention.
  The ocular physiological parameters, including axial length (AL), horizontal and vertical corneal curvature (K1 and K2), were measured using an optical biometer (model IOL Master 700). Each eye was measured three times, and if the difference between any two measurements exceeded 0.05 mm, the process was repeated until the difference was less than this value.An objective examination method was used under non-cycloplegic conditions (i.e., without pupil dilation), utilizing a tabletop automatic refractometer (ISO 10342-2010 Ophthalmic Instruments - Refractometers). The spherical equivalent (SE) was calculated as follows: SE = sphere power + 1/2 cylinder power.

SECONDARY OUTCOMES:
The incidence of myopia. | at baseline, and at the 12th month of the intervention.
  The incidence of myopia is defined as the occurrence of myopia in children who were not myopic at baseline.